CLINICAL TRIAL: NCT02684487
Title: Vitamin D Status in Patients With Severe Sepsis: A Randomized Clinical Trial
Brief Title: Vitamin D Status in Patients With Severe Sepsis
Acronym: ViDISS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left institution. Protocol not submitted to IRB, contract not executed, and study was not done.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ViDISS_temp
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Sepsis; Severe Sepsis; End Organ Damage; Multi Organ Failure
Keywords: vitamin D; vitamin D3; sepsis; severe sepsis; critical illness; ICU
MeSH Terms: conditions — Sepsis; Multiple Organ Failure; Critical Illness | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- vitamin D3 (Active Comparator): Patients will be given single dose of vitamin D3 within 24 hours of new-onset severe sepsis, followed by weekly doses of vitD3 (25,000 IU) up to 90 days to assess clinical outcomes and key biomarkers.
  Interventions: Drug: vitamin D3
- Placebo (Sham Comparator): Patients will be given placebo intervention within 24 hours of new onset severe sepsis followed by or placebo for up to 90 days to assess clinical outcomes and key biomarkers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vitamin D3 — Patients will be given 400,000 IU of vitamin D3 within 24 hours of severe sepsis onset followed by weekly doses of 25,000 IU until 90 days or death, whichever comes first.
  Other Names: cholecalciferol
  Arms: vitamin D3
Drug: Placebo — Patients will be given placebo within 24 hours of severe sepsis onset followed by weekly doses of placebo until 90 days or death, whichever comes first.
  Other Names: sugar pill, sham comparator
  Arms: Placebo

SUMMARY:
Sepsis is a clinical entity that complicates infection. Without early recognition and timely management, it can rapidly progress to severe sepsis, septic shock, and culminate in multiple organ dysfunction syndrome. Forty to 70% of septic patients have low vitamin D status, yet little is known about the impact of vitamin D3 (vitD3) supplementation in this patient population. As such, the investigators propose a randomized, double-blinded, placebo-controlled trial to test the hypothesis that early, rapid correction of low vitamin D status, as an adjunct to established treatment guidelines, will improve clinical outcomes and measurably alter immune profile in patients with severe sepsis.

DETAILED DESCRIPTION:
Sepsis is a clinical entity that complicates infections [1]. Without early recognition and timely management, it can rapidly progress to severe sepsis, septic shock, and culminate in multiple organ dysfunction syndrome. The incidence of severe sepsis is between 300 to 1000 cases per 100,000 persons [2] and is projected to increase annually due to an aging population, increasing burden of chronic disease, and greater use of invasive procedures, chemotherapy, and immunosuppressive agents [3]. Severe sepsis is the leading cause of mortality in critically ill patients, with healthcare costs exceeding $16 billion annually [4]. Despite evolving clinical guidelines for sepsis [5-7], and intense research, only a modest reduction in case fatality rates has been documented over the last two decades [8]. Aside from early administration of antibiotics, there is no effective stand-alone or adjuvant pharmacological intervention to improve survival in patients with severe sepsis.

The degree of immune dysfunction precipitated by an inciting infection is thought to correlate with the severity of sepsis. Recently, key cells of the immune system were shown to express the vitamin D receptor (VDR) [9]. Additionally, macrophages and neutrophils activated through VDR up-regulate expression of endogenous antimicrobial peptides (AMPs) that are active against a broad spectrum of infectious agents [10]. AMPs, influenced by vitamin D status, likely represent an important first-line of defense against microbial invasion. While circulating 25-hydroxyvitamin D (25OHD) is the most abundant vitamin D metabolite [11], under normal circumstances, 85-90% of 25OHD is tightly bound to vitamin D binding protein (DBP) and is unavailable to activate innate immune responses during acute stress [12]. The remaining 10-15% is more readily bioavailable (b25OHD), and is composed of the free and albumin-bound components of 25OHD. Fluid loading, albumin wasting, and increased DBP expression during critical illness may affect 25OHD homeostasis [13].

Low vitamin D status (25OHD <20ng/mL) is associated with increased mortality in critical illness [14]. Forty to 70% of septic patients have low vitamin D status [15-17], yet little is known about the impact of vitamin D3 (vitD3) supplementation in this patient population. As such, the investigators propose a randomized, double-blinded, placebo-controlled trial to test the hypothesis that early, rapid correction of low vitamin D status, as an adjunct to established treatment guidelines, will improve clinical outcomes and measurably alter immune profile in patients with severe sepsis. Patients will be assigned to a single dose of vitD3 (400,000 IU) or placebo (n=300/arm) within 24 hours of new-onset severe sepsis, followed by weekly doses of vitD3 (25,000 IU) or placebo, respectively, up to 90 days to assess clinical outcomes and key biomarkers.

AIM 1: To determine if early administration of vitD3 (vs placebo) improves clinical outcomes in patients with low vitamin D status and severe sepsis. Hypothesis 1a: Early vitD3 decreases 90-day mortality after onset of severe sepsis (Primary Outcome). Hypothesis 1b: Early vitD3 decreases sequential organ failure assessment scores in the first 5 days after onset of severe sepsis. Hypothesis 1c: Early vitD3 decreases non-home discharge rate in those who survive severe sepsis.

AIM 2: To determine if early administration of vitD3 (vs placebo) modulates b25OHD, AMPs, and key cytokines in patients with low vitamin D status and severe sepsis. Hypothesis 2a: Early vitD3 increases b25OHD in the first 5 days after the onset of severe sepsis. Hypothesis 2b: Early vitD3 increases expression of AMPs, cathelicidin (LL-37) and β-defensin (hBD-2). Hypothesis 2c: Early vitD3 decreases pro-inflammatory cytokine (IL-1β, IL-6) and increases anti-immunoparalytic cytokine (IL-10, IFN-γ) expression.

Severe sepsis is a significant public health problem with limited treatment options. A 2010 NIH workshop on sepsis identified deep gaps in understanding innate host immune responses in sepsis and emphasized the need for novel therapies [18]. The proposed trial is well powered to investigate whether immunomodulation with vitD3 improves survival after severe sepsis. By optimizing endogenous host responses to infection, the investigators anticipate that vitD3 supplementation will augment the life-saving impact of current therapies for severe sepsis. Moreover, the investigators will investigate several vitamin D-related biomarkers, which may identify future therapeutic targets. The trial will be performed by a highly-experienced team that includes experts in vitamin D, sepsis, critical care, and clinical trials; they have successfully carried out several clinical studies of vitamin D in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to <80 years
* Admitted to 1 of 4 participating ICUs
* Meet criteria for new-onset severe sepsis* within past 12 hours

Exclusion Criteria:

* Age ≥80 years
* Not anticipated to survive ≥48 hours
* Inability to obtain informed consent from patient/suitable proxy within 22 hours of new-onset severe sepsis
* Comfort measures, hospice, or palliative care status
* Documented adverse reaction to vitamin D supplementation
* Inability to tolerate enteral feeds/medications
* Renal stones within past year
* Hypercalcemia within past year
* Baseline serum calcium ≥10.5 mg/dL
* Established diagnosis of medical condition associated with high risk of hypercalcemia (e.g. metastatic cancer, sarcoidosis, multiple myeloma, primary hyperparathyroidism)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
90 day mortality | 90 day mortality
  90 day mortality will be assessed in patients included in the study

SECONDARY OUTCOMES:
Serum b25OHD: Baseline serum b25OHD and serum b25OHD after intervention, until hospital day 5 | 24h of severe sepsis onset until hospital day 5
  b25 OHD will be measured in the first 5 days after the onset of severe sepsis
Serum measurement of AMPs, cathelicidin, and B-defensin: Baseline serum AMPs, cathelicidin, and B-defensin and AMPs, cathelicidin, and B-defensin after intervention, until hospital day 5 | 24h of severe sepsis onset until hospital day 5
  AMPs, Cathelicidin and B-defensin will be measured in the first 5 days after the onset of severe sepsis
Serum measurement of cytokines: Baseline serum cytokines and serum cytokines after intervention, until hospital day 5 | 24h of severe sepsis onset until hospital day 5
  IL1B, IL-6, IL-10 and IFN-y will be measured in the first 5 days after the onset of severe sepsis
sequential organ failure assessment scores in the first 5 day after severe sepsis onset | 24h of severe sepsis onset until hospital day 5
  SOFA scores will be taken within the first 5 days of onset of severe sepsis in patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A Quraishi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes